CLINICAL TRIAL: NCT01500161
Title: A Phase II Study Of Pooled Unrelated Donor Umbilical Cord Blood (UCB) Transplant For Patients With Hematologic Malignancies Needing Allogeneic Stem Cell Transplant But Do Not Have A Related HLA-Matched Donor
Brief Title: Pooled Unrelated Donor Umbilical Cord Blood Transplant For Hematologic Malignancy Needing Allogeneic Stem Cell Transplant Without Related HLA-Match
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accruals
Sponsor: Texas Oncology Cancer Center (Industry)
Responsible Party: Principal Investigator, Seah Lim M.D., Principle Investigator, Texas Oncology Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1127920
Record Dates: First submitted 2011-11-18; First posted 2011-12-28 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Hodgkins Disease; Non-Hodgkins Lymphoma; Aplastic Anemia; Multiple Myeloma; Myelodysplastic Syndrome
Keywords: Leukemia; Lymphoma; Myeloma; Aplastic Anemia; Myelodysplasia; AML; ALL; CLL; CML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Lymphoma, Non-Hodgkin; Anemia, Aplastic; Multiple Myeloma; Myelodysplastic Syndromes; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Anemia, Refractory, with Excess of Blasts | interventions — Busulfan; Clofarabine; fludarabine; Melphalan; Carmustine; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): The following conditioning regimens will be used, depending on the underlying hematologic malignancies. Conditioning regimens with Busulfan/clofarabine and with fludarabine/melphalan will be used for all patients except those with Non-Hodgkin's lymphoma when the conditioning regimen of BCNU, Etoposide, ARA-C and Melphalan will be used.
  Interventions: Drug: Busulfan; Drug: Clofarabine; Drug: Fludarabine; Drug: Melphalan; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine

INTERVENTIONS:
Drug: Busulfan — Busulfan 3.2 mg/kg/day intravenously on days -7, -6, -5 and -4(for non-NHL patients patients who get Clofarabine regimen)
Drug: Clofarabine — Clofarabine intravenously 40 mg/m2/day on days -7, -6, -5, -4 and -3(for non-NHL patients patients who get Busulfan regimen)
Drug: Fludarabine — Fludarabine 30 mg/kg/day intravenously on days -7, -6, -5, -4 and -3 (for non-NHL patients who receive Melphalan containing regimen)
Drug: Melphalan — Melphalan intravenously 140 mg/m2/day on day -3 (only for non-NHL patients who receive Fludarabine OR for all NHL regimens)
Drug: Carmustine — BCNU(Carmustine)300 mg/m2 intravenously on day -7 (for NHL patients only)
Drug: Etoposide — Etoposide 300 mg/m2/day intravenously on days -6, -5, -4 and -3 (for NHL patients only)
Drug: Cytarabine — ARA-C(Cytarabine) 100 mg/m2/day on days -6, -5, -4 and -3 (for NHL patients only)

SUMMARY:
The purpose of this study is to evaluate the multi-lineage hematopoietic chimerism for unrelated umbilical cord blood (UCB) grafts pooled from two to three cord blood units. Also to evaluate the toxicity, and antitumor responses of pooled unrelated UCB transplants.

DETAILED DESCRIPTION:
Hematopoietic stem cell (HSC) transplantation, using human HLA-matched sibling or unrelated bone marrow or peripheral blood stem cell donor, has been used successfully to treat patients with high-risk or relapsed hematologic malignancies. However, use of this therapy has been limited by availability of fully HLA-matched donors, despite the increasing size of unrelated donor registries. For those transplanted with unrelated donor marrow stem cells, increased HLA disparity adversely affects survival due to increased risks of severe acute and chronic graft-versus-host disease (GVHD) and opportunistic infection. Only young recipients are able to tolerate a single HLA-A, B, DRB1 mismatch in this setting (1-3). To potentially extend the donor pool, UCB has been used as an alternative source of HSC. Since the first unrelated donor UCB transplant in 1993, UCB transplants have been performed worldwide. It has been found to produce outcome comparable to those from matched unrelated HSC in patients with hematologic malignancies (4). It has been shown that cryopreserved unrelated UCB from 0 to 3 HLA-A, B, DRB1-mismatched donors contains sufficient HSC to engraft most pediatrics and some adult patients (5-10). Unfortunately, the use of UCB transplant is limited by the small number of HSC in each of the cord blood unit. This is particularly a problem for adult patients. It is now possible to pool UBC so that adequate cell numbers are available for adult transplant (11). UBC is rapidly availability and has very low rate of contamination with herpes group viruses. UCB transplant results in a low incidence of both severe acute GVHD and extensive chronic GVHD, despite the use of grafts with substantial donor-recipient HLA disparity (5-10).

The following conditioning regimens will be used, depending on the underlying hematologic malignancies. Conditioning regimens with Busulfan/clofarabine and with fludarabine/melphalan will be used for all patients except those with Non-Hodgkin's lymphoma when the conditioning regimen of BCNU, Etoposide, ARA-C and Melphalan will be used. GVHD prophylaxis of oral tacrolimus will be used, depending on the development of GVHD and the clinical conditions of the patients, tacrolimus may be tapered and discontinued by six months after transplant. The hematopoietic stem cells from the donors will be infused within 48-72 hours of completing the chemotherapy. The patients will receive supportive care as indicated including antibiotics, antivirals, antifungals, anti-seizure, anti-emetic medications and other medications as necessary. In addition patients will receive irradiated blood products for support as necessary.CMV negative recipient transplant will receive only CMV- blood products. Neutrophil engraftment will be defined as the day on which the ANC rises to > 500 cells/ml for two consecutive days. Platelet engraftment will be defined as the first day on which the platelet count rises to > 20,000/ml over a 7-day interval without transfusion support.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 65 years with hematologic malignancies needing stem cell transplant but do not have HLA-matched sibling donor. Patients with the following diagnosis will be included:

  * AML in first or subsequent complete or partial remissions
  * ALL in first or subsequent complete or partial remissions
  * CLL in second remission or more advanced disease
  * CML who has failed tyrosine kinase inhibitors
  * Hodgkin's disease who relapse after autologous transplant
  * Non-Hodgkin's lymphoma who relapse after autologous transplant or NK-cell lymphoma in CR1
  * Aplastic anemia patients
  * Multiple myeloma in second remission or moer advanced disease, including those who have failed an autologous transplant
  * Myelodysplastic syndrome in first or subsequent complete or partial remission
* Patients must have 6/6, 5/6 or 4/6 molecular matches from unrelated UCB donors. Matching will be done for A, B, and DR. Matching at DR will be confirmed by molecular typing.
* Patients must be documented to be HIV negative. Screening must have been performed within previous 6 months.
* Patients must be able to give written consent.

Exclusion Criteria:

* Patient is excluded if all of the Inclusion criteria above isn't met.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
evaluate the multi-lineage hematopoietic chimerism for unrelated UCB grafts pooled from two to three cord blood units | Will be tested after granulocyte engraftment - which will happen at an average of 28 days post-transpant
  Blood will be obtained for DNA preparation for VNTR chimerism study post transplant after time of engraftment, which will happen at an average of 28 days post-trasplant.

SECONDARY OUTCOMES:
evaluate the antitumor responses of pooled UCB transplant | Disease staged at baseline, then disease status re-assessed at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that every 6 months post-transplant
  Baseline - All patients will have a detailed history and physical examination, CBC, complete biochemical profile and full staging procedure appropriate for the underlying disease.
  Post Transplant Evaluation- Disease status will be assessed prior to discharge, again at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that every 6 months.The following data will be collected: hematologic recovery, and grade and tumor responses and duration of response.
Number of participants that develop Graft Versus Host Disease after pooled UCB transplant | Patients will be assessed weekly during first 28 days then re-assessed at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that every 6 months post-transplant.
  Baseline - All patients will have a detailed history and physical examination, CBC, complete biochemical profile.
  Post Transplant Evaluation- Patient will be evaluated prior to discharge,then weekly for first 28 days then re-assessed at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that every 6 months. The following data will be collected: Patient will be assessed for any ongoing adverse events, and CBC's and biochemical profile's will be performed.
The Infection rate seen in the participants who received a pooled UCB transplant | Patients will be assessed weekly during first 28 days then re-assessed at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that every 6 months post-transplant.
  Baseline - All patients will have a detailed history and physical examination, CBC, complete biochemical profile.
  Post Transplant Evaluation- Patient will be evaluated prior to discharge,then weekly for first 28 days then re-assessed at 6 weeks, 3 months, 6 months, 9 months, 12 months and after that every 6 months. The following data will be collected: Patient will be assessed for any ongoing adverse events, and CBC's and biochemical profile's will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Seah Lim, MD, Principal Investigator — Texas Oncology - Amarillo,TX
Locations (1):
- Texas Oncology, Amarillo, Texas, United States

REFERENCES:
- [Background] Balduzzi A, Gooley T, Anasetti C, Sanders JE, Martin PJ, Petersdorf EW, Appelbaum FR, Buckner CD, Matthews D, Storb R, Sullivan KM, Hansen JA. Unrelated donor marrow transplantation in children. Blood. 1995 Oct 15;86(8):3247-56. PMID 7579422
- [Background] Petersdorf EW, Longton GM, Anasetti C, Martin PJ, Mickelson EM, Smith AG, Hansen JA. The significance of HLA-DRB1 matching on clinical outcome after HLA-A, B, DR identical unrelated donor marrow transplantation. Blood. 1995 Aug 15;86(4):1606-13. PMID 7632970
- [Background] Laughlin MJ, Barker J, Bambach B, Koc ON, Rizzieri DA, Wagner JE, Gerson SL, Lazarus HM, Cairo M, Stevens CE, Rubinstein P, Kurtzberg J. Hematopoietic engraftment and survival in adult recipients of umbilical-cord blood from unrelated donors. N Engl J Med. 2001 Jun 14;344(24):1815-22. doi: 10.1056/NEJM200106143442402. PMID 11407342
- [Background] Wagner JE, Kernan NA, Steinbuch M, Broxmeyer HE, Gluckman E. Allogeneic sibling umbilical-cord-blood transplantation in children with malignant and non-malignant disease. Lancet. 1995 Jul 22;346(8969):214-9. doi: 10.1016/s0140-6736(95)91268-1. PMID 7616801
- [Background] Wagner JE, Rosenthal J, Sweetman R, Shu XO, Davies SM, Ramsay NK, McGlave PB, Sender L, Cairo MS. Successful transplantation of HLA-matched and HLA-mismatched umbilical cord blood from unrelated donors: analysis of engraftment and acute graft-versus-host disease. Blood. 1996 Aug 1;88(3):795-802. PMID 8704232
- [Background] Kurtzberg J, Laughlin M, Graham ML, Smith C, Olson JF, Halperin EC, Ciocci G, Carrier C, Stevens CE, Rubinstein P. Placental blood as a source of hematopoietic stem cells for transplantation into unrelated recipients. N Engl J Med. 1996 Jul 18;335(3):157-66. doi: 10.1056/NEJM199607183350303. PMID 8657213
- [Background] Gluckman E, Rocha V, Boyer-Chammard A, Locatelli F, Arcese W, Pasquini R, Ortega J, Souillet G, Ferreira E, Laporte JP, Fernandez M, Chastang C. Outcome of cord-blood transplantation from related and unrelated donors. Eurocord Transplant Group and the European Blood and Marrow Transplantation Group. N Engl J Med. 1997 Aug 7;337(6):373-81. doi: 10.1056/NEJM199708073370602. PMID 9241126
- [Background] Rubinstein P, Carrier C, Scaradavou A, Kurtzberg J, Adamson J, Migliaccio AR, Berkowitz RL, Cabbad M, Dobrila NL, Taylor PE, Rosenfield RE, Stevens CE. Outcomes among 562 recipients of placental-blood transplants from unrelated donors. N Engl J Med. 1998 Nov 26;339(22):1565-77. doi: 10.1056/NEJM199811263392201. PMID 9828244